CLINICAL TRIAL: NCT05315817
Title: Safety and Performance Evaluation of multiPlus Dialysate During CRRT
Acronym: multiPlus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal reasons
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRRT-CVVHD(F)/MP-01-D
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Acute Kidney Injury
Keywords: Renal replacement therapy; Acute kidney injury; Haemodialysis; Haemodiafiltration
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Prospective, non-comparative, multi-centre, open-label, interventional, post market clinical follow-up (PMCF) study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multiPlus dialysate (Experimental): Treatment of acute kidney injury patients either with continuous veno-venous haemodialysis (CVVHD) or continuous veno-venous haemodiafiltration (CVVHDF) using the multiPlus dialysate.
  Interventions: Device: multiPlus dialysate

INTERVENTIONS:
Device: multiPlus dialysate — Treatment of acute kidney injury patients either with continuous veno-venous haemodialysis (CVVHD) or continuous veno-venous haemodiafiltration (CVVHDF) using the multiPlus dialysate.

SUMMARY:
Assessment of the performance of multiPlus dialysate based on the serum creatinine removal 6 hours (360 min) after start of continuous veno-venous haemodialysis/ haemodiafiltration [CVVHD(F)].

multiPlus is a phosphate-containing dialysis solution for the use in continuous renal replacement therapy (CRRT) during acute kidney injury (AKI).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form by investigator and by

  * a) the study patient: if patient is able to consent
  * b) the legal representative: if patient is unable to consent:
  * c) an independent consultant: in case of emergency
* if c) either legal representative or study patient, whichever can be done sooner, should be informed by the investigator as soon as possible. If the informed consent has been obtained by the legal representative (b or emergency scenario) informed consent to continue the participation in the clinical investigation shall be obtained from the subject as soon as he or she is capable of giving informed consent (According to the MDR - Article 68 - Clinical investigations in emergency situations)
* Minimum age of 18 years
* Ability to understand the nature and requirements of the study (if patient is conscious)

Study specific:

* Body weight greater than 40 kg
* Acute Kidney Injury (AKI) with clinical indication for CVVHD/CVVHDF
* Vascular access allowing blood flow of min 50mL/min
* Estimated life expectancy greater than 3 days

Exclusion Criteria:

* Any conditions which could interfere with the patient's ability to comply with the study
* In case of female patients: pregnancy (negative pregnancy test for women below 55 years) or lactation period
* Participation in an interventional clinical study during the preceding 30 days
* Previous participation in the same study
* SARS-CoV 2 positive

Study specific

* Hyperphosphataemia (>4.5 mg/dL)
* Hypersensitivity to heparin or known history of heparin induced thrombocytopenia (HIT Type II)
* Uncontrolled bleeding and coagulation disorders
* Decision to limit therapeutic interventions
* Advanced malignancy (not including myeloma)
* Dementia (if definitely not an acute confusional state from uraemia or other acute illness)
* Advanced cirrhosis with encephalopathy in the absence of possible liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Serum creatinine removal | 360 min after start
  The primary variable of this clinical investigation is serum creatinine removal (arterial pre-filter sample taking) assessed 6 hours (360 min) after start of CVVHD(F).

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Borger, Prof Dr, Principal Investigator — Helios Health Institute GmbH
Locations (1):
- Leipzig Heart Institute GmbH, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No